CLINICAL TRIAL: NCT06858982
Title: The Polish Mother's Memorial Hospital Research Institute Pitavastatin Registry
Brief Title: PMMHRI-Pitavastatin Registry
Status: Recruiting | Type: Observational
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PMMHRI-Pitavastatin Registry
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; pitavastatin
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The PMMHRI-Pitavastatin Registry is a non-interventional, single-center registry conducted at the Polish Mother's Memorial Hospital Research Institute (PMMHRI). Established in January 2024, the registry enrolls all patients from the Department of Cardiology and Adult Congenital Heart Diseases, the Department of Endocrinology, as well as outpatient cardiology and endocrinology clinics who are prescribed pitavastatin.

DETAILED DESCRIPTION:
The PMMHRI-Pitavastatin Registry is a non-interventional, single-center registry conducted at the Polish Mother's Memorial Hospital Research Institute (PMMHRI), the second-largest supra-regional hospital in Poland. The registry was initiated in January 2024 to systematically collect real-world data on patients prescribed pitavastatin, aiming to assess its effectiveness, safety, and impact on lipid and cardiovascular risk management.

The registry has included all patients from the Departments of Cardiology and Endocrinology, as well as outpatient cardiology and endocrinology clinics, who have been prescribed pitavastatin. The inclusion of a broad patient population allows for a comprehensive evaluation of treatment patterns and outcomes in routine clinical practice.

Patient data are extracted from electronic medical records and include:

Demographic parameters (age, sex, BMI, etc.) Relevant comorbidities (e.g., hypertension, diabetes, chronic kidney disease) Concomitant medications, including: Lipid-lowering therapy status (monotherapy vs. combination therapy), Anticoagulation status Lifestyle factors, such as smoking status Post hoc calculated cardiovascular risk scores, to stratify patients based on their predicted risk of major adverse cardiovascular events (MACE) Laboratory parameters, including lipid profiles, inflammatory markers, and metabolic indicators.

ELIGIBILITY:
Inclusion Criteria:

* patient takling pitavastatin based on the 2021 Polish Lipid Guidelines

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Department of Cardiology and Adult Congenital Heart Diseases, Department of Endocrinology, and outpatient cardiology and endocrinology clinics who is taking pitavastatin.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Patient's characteristic. | 5 years
  Characteristic of patients treated with pitavastatin among the Polish population.

CONTACTS AND LOCATIONS:
Locations (1):
- Polish Mother's Memorial Hospital Research Institute, Lodz, Poland